CLINICAL TRIAL: NCT06309212
Title: Assessing the Impact of COVID-19 on HMPV Incidence and Severity Among Adults
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-20/687
Record Dates: First submitted 2024-03-12; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: The Prevalance of HMPV After COVID-19 Pandemic; The Importance of Accurate Diagnosis for HPMV
Keywords: Adults; Human metapneumovirus; Post-COVID-19 era; Prevalence; Underestimated Virus
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-COVID period: January 2016 to January 2020
  Interventions: Other: Observation
- Post-COVID period: January 2021 to September 2023
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Analyse of data from adults with respiratory tract infections who were tested for various respiratory viruses using a multiplex PCR assay

SUMMARY:
Human metapneumovirus (HMPV) is primarily recognized as a childhood pathogen, but its impact on adults remains largely underestimated. This study investigates the prevalence, clinical characteristics, and post-COVID-19 trends of HMPV infection among adults in Istanbul, Turkey.

DETAILED DESCRIPTION:
Human metapneumovirus (HMPV) is primarily recognized as a childhood pathogen, but its impact on adults remains largely underestimated. This study investigates the prevalence, clinical characteristics, and post-COVID-19 trends of HMPV infection among adults in Istanbul, Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years
* Patients with acute respiratory tract infection symptoms
* Patients who underwent multiplex PCR testing for respiratory viruses

Exclusion Criteria:

* Patients for whom no respiratory viral panel test was conducted

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study examined adults with acute respiratory tract infections in Istanbul, Turkey. Patients admitted between 2016-2020 (pre-COVID) and 2021-2023 (post-COVID) underwent multiplex PCR testing for various respiratory viruses, with a focus on human metapneumovirus. The study aimed to assess the prevalence of HMPV infection in adults and its potential change after the COVID-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 2197 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of HMPV infection in adults pre- and post-COVID-19 pandemic | Between 2016-2020 (pre-COVID) and 2021-2023 (post-COVID)
  Analyse of data from adults with respiratory tract infections who were tested for various respiratory viruses using a multiplex PCR assay

SECONDARY OUTCOMES:
Comparison of HMPV with other respiratory viruses in adults | Between 2016-2020 (pre-COVID) and 2021-2023 (post-COVID)
  Analyse of data from adults with respiratory tract infections who were tested for various respiratory viruses using a multiplex PCR assay

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Niederman MS, Torres A. Respiratory infections. Eur Respir Rev. 2022 Oct 19;31(166):220150. doi: 10.1183/16000617.0150-2022. Print 2022 Dec 31. PMID 36261160
- [Background] Haas LE, Thijsen SF, van Elden L, Heemstra KA. Human metapneumovirus in adults. Viruses. 2013 Jan 8;5(1):87-110. doi: 10.3390/v5010087. PMID 23299785
- [Background] Boivin G, De Serres G, Hamelin ME, Cote S, Argouin M, Tremblay G, Maranda-Aubut R, Sauvageau C, Ouakki M, Boulianne N, Couture C. An outbreak of severe respiratory tract infection due to human metapneumovirus in a long-term care facility. Clin Infect Dis. 2007 May 1;44(9):1152-8. doi: 10.1086/513204. Epub 2007 Mar 28. PMID 17407031
- [Background] Chow EJ, Uyeki TM, Chu HY. The effects of the COVID-19 pandemic on community respiratory virus activity. Nat Rev Microbiol. 2023 Mar;21(3):195-210. doi: 10.1038/s41579-022-00807-9. Epub 2022 Oct 17. PMID 36253478
- [Background] Pearson V. Case studies. Baton Rouge puts community first. Trustee. 1995 May;48(5):24-6. No abstract available. PMID 10142898